CLINICAL TRIAL: NCT03813862
Title: OPERA Longitudinal Observational Database in the Study of Chronic Diseases, Treatments and Outcomes
Brief Title: Observational Pharmaco-Epidemiology Research & Analysis
Acronym: OPERA
Status: Recruiting | Type: Observational
Sponsor: Epividian (Industry)
Responsible Party: Sponsor
Other Study IDs: Pro00023648
Record Dates: First submitted 2019-01-11; First posted 2019-01-23 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2025-02

CONDITIONS: Chronic Disease; HIV/AIDS; Liver Diseases; Inflammatory Bowel Diseases; Cardiovascular Diseases; Rheumatic Diseases; Neurodegenerative Diseases
MeSH Terms: conditions — Chronic Disease; Acquired Immunodeficiency Syndrome; Liver Diseases; Inflammatory Bowel Diseases; Cardiovascular Diseases; Rheumatic Diseases; Neurodegenerative Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: Non-interventional (observational only)

SUMMARY:
Greater advances are needed in two separate but related areas in healthcare: 1) the Clinical Decision Support Systems that complement the EHR use in support of routine patient care, population management and disease management; and 2) the use of the point-of-care observational data from the provider-patient encounter that support realworld medical research and healthcare quality measure assessment. Real-world evaluations of treatments of chronic diseases in the context of comorbid conditions and special populations (minorities, women, mentally ill, and those with addiction) are limited. The purpose of the OPERA database is to help address this unmet need in clinical research.

DETAILED DESCRIPTION:
Objectives of OPERA

1. To research numerous chronic diseases (HIV, HCV, HBV currently and IBD and RA in the near future, with others as identified for further consideration) utilizing the OPERA® longitudinal database that consists of de-identified EHR data from numerous clinical practices in a variety of settings (e.g. solo practitioners, small groups, and hospitals). Research will be ongoing and yield numerous individual analyses and reports that are authored by epidemiologists, practicing physicians, pharmaco-economists, and other researchers and will target scientific conferences and peer-reviewed medical journals for dissemination.
2. To use epidemiological, statistical, and data analysis methods and related research findings to deliver a sophisticated healthcare analytics reporting solution (CHORUS™) to clinicians.†
3. To enhance patient population management as well as disease management capabilities of the practicing physician.
4. To provide anonymous, nation-wide benchmarking of quality measures and key performance indicators (KPI) for medical clinics.
5. To enhance patient engagement with their physicians to deliver better health outcomes.
6. To evaluate whether engagement in care by patients with their physicians results in better outcomes for patients with chronic illness.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are treated in the practices who enroll and participate in the study
* Patients whose treatment is documented in the practice's electronic health record system

Exclusion Criteria:

* Patients who opt out of OPERA

Min Age: 0 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The patient population includes a diverse group of individuals treated in ambulatory practice with a focus on those living with chronic disease.
Sampling Method: Probability Sample
Enrollment: 2000000 (Estimated)
Dates: Start 2013-12-01 (Actual); Primary Completion 2035-11 (Estimated); Study Completion 2035-11 (Estimated)

PRIMARY OUTCOMES:
Virologic response to therapy | 1 year
  HIV-1 PCR laboratory value ("viral load") quantifies the amount of HIV-1 copies in plasma per mL. The baseline viral load is compared to viral load after 1 year of antiretroviral therapy.

CONTACTS AND LOCATIONS:
Locations (1):
- Epividian, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No